CLINICAL TRIAL: NCT06583330
Title: A Multicenter, Open-Label, Non-Inferiority Randomized Controlled Trial of Postoperative VTE Prevention in Chinese Patients After Colorectal Cancer Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BFH-VTE
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Surgery; VTE (Venous Thromboembolism)
MeSH Terms: conditions — Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight; Dalteparin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Low molecular weight heparin should be initiated for drug prevention within 24 hours after surgery, with a preventive course of 14 days
  Interventions: Drug: Low Molecular Weight Heparin (dalteparin)
- control arm (Active Comparator): All patients should initiate low molecular weight heparin for drug prophylaxis within 24 hours after surgery, with a prophylaxis course of 28 days
  Interventions: Drug: Low Molecular Weight Heparin (dalteparin)

INTERVENTIONS:
Drug: Low Molecular Weight Heparin (dalteparin) — All patients initiated low molecular weight heparin for drug prevention within 24 hours after surgery. The prevention course for the experimental group patients was 14 days, while the prevention course for the control group patients was 28 days. Low molecular weight heparin is administered subcutaneously once daily at a dose of 0.3ml.

SUMMARY:
research objective

1. Optimize VTE prevention management after CRC surgery.
2. Improve the prevention and treatment level of VTE in current perioperative patients.
3. Reduce the social burden of VTE related diseases.

Participants will:

1. start low molecular weight heparin prophylaxis within 24 hours post-surgery.
2. The prophylactic regimen for the experimental group lasted 14 days, while the control group received it for 28 days. Low molecular weight heparin is given subcutaneously at a dose of 0.3ml once daily.
3. atients underwent lower limb color Doppler ultrasound on postoperative days 7 ± 2, 14 ± 3, and 28 ± 5, which included screening for thrombosis in the proximal deep veins (femoral, popliteal), distal deep veins (posterior tibial, fibular, and muscular veins), and their perforating branches.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years old; Diagnosed with colorectal cancer and undergoing curative, palliative, or other limited surgeries (laparoscopic or open surgery), with an estimated surgery time of>45 minutes; Expected postoperative survival>6 months; Expected Caprini score of ≥ 5 on the first day after surgery; The patient agrees to the research plan and signs an informed consent form.

Exclusion Criteria:

* Renal dysfunction (CrCl<30 mL/min) or liver dysfunction (ALT>3 times the upper limit of normal); Known allergies to LMWH, anesthetics, or contrast agents; There is a systemic bleeding disorder or bleeding tendency, such as active peptic ulcer, uncontrolled hypertension, cerebral thrombosis within 6 months, cerebral hemorrhage, or a history of neurosurgical surgery; Known brain metastases, endocarditis, or previous heparin induced thrombocytopenia; VTE occurred within 3 months before surgery; Use heparin or oral anticoagulant therapy within 5 days before surgery; Pregnant or lactating women; Pregnant or lactating women; Any conditions that researcher determines the subject not suitable for anticoagulant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1448 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
VTE events, including deep vein thrombosis (DVT) and pulmonary thromboembolism (PE). | From enrollment to the end of treatment at 4 weeks